CLINICAL TRIAL: NCT07161830
Title: Evaluation of the Efficacy of Omeza® Complete Matrix in the Healing of Chronic Diabetic Foot Ulcers: A Randomized Controlled Multicenter Crossover Trial
Brief Title: Evaluating the Efficacy of OCM™ (Omeza® Complete Matrix) in the Treatment of Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Omeza, LLC (Industry)
Collaborators: SygNola, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ocdiam
Record Dates: First submitted 2025-08-27; First posted 2025-09-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Chronic Wounds; Wound Medicine
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The subject will be randomized to one of the following treatments:
  * Standard of care
  * OCM in addition to standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- OCM + SOC (Experimental): Omeza® Complete Matrix (OCM™) is a wound care matrix comprised of hydrolyzed fish collagen derived from whitefish skin
  Interventions: Device: Omeza® Complete Matrix
- Standard of Care (Active Comparator): Surgical sharp debridement, offloading (TCC gold standard, fixed ankle-walker alternative), and proper moisture balance
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Omeza® Complete Matrix — OCM Application, Surgical sharp debridement, offloading (TCC gold standard, fixed ankle-walker alternative), and proper moisture balance
  Other Names: OCM
  Arms: OCM + SOC
Other: Standard of Care — Surgical sharp debridement, offloading (TCC gold standard, fixed ankle-walker alternative), and proper moisture balance
  Other Names: SOC
  Arms: Standard of Care

SUMMARY:
This study aims to compare two treatment approaches for diabetic foot ulcers (DFUs): the standard of care (SOC) alone versus SOC combined with OCM. Researchers will evaluate whether adding OCM increases the likelihood of ulcers healing completely by the end of the trial period.

DETAILED DESCRIPTION:
This research will take place across multiple medical centers, where both researchers and participants will know which treatment is being used (open label). Patients who agree to participate and meet the study requirements during screening will be randomly assigned to one of two groups: either standard of care (SOC) alone, or SOC plus OCM. The study includes a crossover component for subjects in the SOC arm. At treatment visit 13 (approximately 84 days post-randomization), SOC arm subjects not having achieved complete wound closure, and still meeting the inclusion/exclusion criteria, are eligible to cross over to the IP arm (SOC plus OCM). Crossover subjects will begin IP arm treatment with weekly OCM applications for up to 12 treatment visits. The subject will continue follow-up per the original schedule. As this is a post-marketing study, it will gather information regarding the efficacy of treatment while also supporting insurance reimbursement decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Subject has a medical diagnosis of Type I or Type II Diabetes Mellitus requiring oral or glycemic control and/or insulin replacement therapy
3. Subject has a diabetic foot ulcer present for 4 weeks or greater (documented in medical record), and less than 12 months duration if being treated with continuous SOC
4. Subject has a diabetic foot ulcer with a historical wound measurement showing less than 25% healing in 14 days prior to screening
5. Subject has a diabetic foot ulcer with screening wound measurement showing less than 25% healing in 14 days prior to randomization
6. Subject has a diabetic foot ulcer of Wagner grade 1, 2, or 3 without infection or clinically visible exposed bone. Wagner 3 is acceptable if the diagnosis is acute osteomyelitis and the subject has successfully completed IV antibiotic treatment prior to screening.
7. Index ulcer is a minimum of 0.7cm2 and a maximum of 25cm2 at first treatment visit
8. Diabetic foot ulcer is being treated with offloading therapy for 14 days prior to randomization
9. Adequate circulation of ulcer demonstrated by an ABI of >0.7 and <1.3, or TBI of >0.6 within 30 days prior to randomization OR an arterial ultrasound noted with patent circulation and without significant stenosis 90 days prior to randomization.
10. Index ulcer is free of infection prior to randomization and during screening phase. Infection must be adequately treated and controlled as defined by Infectious Disease Society of America (IDSA) Guidelines PEDIS Grade 1.
11. Index ulcer is free of necrotic debris prior to OCMTM application
12. Female subjects of childbearing potential having a negative pregnancy test prior to randomization
13. Subject is able and willing to follow the protocol requirements
14. Subject had signed informed consent
15. If 2 or more ulcers are present, the ulcers must be separated by at least 2 cm

Exclusion Criteria:

1. Subject has a known life expectance of <1 year
2. Subject is unable to comply with protocol treatment
3. Subject has major uncontrolled medical disorders in the opinion of the investigator, such as serious cardiovascular, renal, liver, pulmonary, autoimmune, palliative care, or inherited blood disorders that may affect wound healing
4. Subject actively being treated for malignant disease or history of malignancy or radiation therapy at the site of wound
5. Subject has comorbid conditions that may compromise subject safety in the opinion of the investigator
6. Known contraindications to Acellular matrices
7. Concurrent participation in alternative clinical trial that involves investigational drug or device interfering with wound treatment and/or healing
8. Subject is pregnant or breastfeeding
9. Subject with history of immunosuppressant treatment (systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or topical steroid application to the ulcer surface for >2 weeks duration within 30 days prior to randomization; or anticipated use of the above during the course of the study
10. Wound previously treated with CAMPs, tissue engineered, or scaffold materials within 30 days prior to randomization
11. Diabetic foot ulcer of Wagner 3 grade with active acute infection that has not completed IV antibiotic treatment, or Wagner 3 grade with chronic refractory osteomyelitis
12. Wound depth with visible exposed bone
13. HBOT within 14 days prior to randomization
14. Revascularization surgery on the index ulcer leg within 30 days of screening phase
15. Index ulcer suspicious of neoplasm in the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | 1-12 weeks
  The primary endpoint will be the percentage of target ulcers that achieve complete wound closure within 12 weeks.

SECONDARY OUTCOMES:
Percentage Wound Area Change | 1-12 weeks
  The percentage change in wound area from TV-1 to TV-13 will be measured weekly using digital photographic planimetry and physical examination.
Pain Assessment | 1-12 weeks
  Change in pain associated with the target ulcer will be assessed using the Numeric Pain Rating Scale throughout the study. The Numeric Pain Rating Scale is measured between 0-10. 0 being no pain at all and 10 being the worst pain.

OTHER OUTCOMES:
Hemoglobin A1c | 1-16 weeks
  Incidence of wound closure vs HbA1c >10, 12, 15
Time to Closure | 1-12 weeks
  Average number of grafts/weeks used to achieve wound closure
Follow-Up Closure | 2-weeks
  Number of wounds that re-opened during the 2-week follow-up
Adverse Events and Serious Adverse Events | 1-16 weeks
  The number and nature of adverse events (AEs) and serious adverse events (SAEs) occurring during the study will be tracked and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Ferguson, DNP, Study Director — SygNola, LLC
Locations (3):
- United States (3):
  - MedCentris of Denham Springs, Denham Springs, Louisiana
  - MedCentris of Leesville, Leesville, Louisiana
  - MedCentris of Southaven, Southaven, Mississippi